CLINICAL TRIAL: NCT06758401
Title: AN OPEN-LABEL, RANDOMIZED, CONTROLLED PHASE 3 STUDY OF SIGVOTATUG VEDOTIN IN COMBINATION WITH PEMBROLIZUMAB COMPARED WITH PEMBROLIZUMAB MONOTHERAPY AS FIRST-LINE TREATMENT IN PARTICIPANTS WITH PD-L1 HIGH (≥50% OF TUMOR CELLS EXPRESSING PD-L1), LOCALLY ADVANCED, UNRESECTABLE, OR METASTATIC NON-SMALL CELL LUNG CANCER (BE6A LUNG-02)
Brief Title: This is a Study to Learn About How the Combination of the Study Medicines Sigvotatug Vedotin Plus Pembrolizumab Works in People With Non-small Cell Lung Cancer With High Levels of PD-L1.
Acronym: Be6A Lung-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C5751003; 2024-517968-36-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; Carcinoma, Non-Small-Cell Lung (NSCLC)
Keywords: Lung Cancer; Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sigvotatug Vedotin with Pembrolizumab (Experimental): Participants will receive Sigvotatug Vedotin, administered as an IV infusion and pembrolizumab, administered as an IV infusion.
  Interventions: Drug: Sigvotatug Vedotin; Drug: Pembrolizumab
- Pembrolizumab Monotherapy (Active Comparator): Participants will receive pembrolizumab, administered as an IV infusion.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sigvotatug Vedotin — MMAE-Antibody Drug Conjugate targeting Integrin Beta-6
  Arms: Sigvotatug Vedotin with Pembrolizumab
Drug: Pembrolizumab — Anti-PD-(L)1

SUMMARY:
The purpose of the study is to compare how the new combination treatment (Sigvotatug Vedotin plus pembrolizumab) works compared to pembrolizumab alone in patients with non-small cell lung cancer (NSCLC) with high levels of PD-L1. This is a protein that acts as a kind of "brake" to keep the body's immune responses under control.

The study is seeking for participants who:

* Are confirmed to have NSCLC (Stage 3 or 4).
* Have PD-L1 levels in more than 50% of the cancer cells.

All participants in this study will receive pembrolizumab at the study clinic once every 6 weeks as an intravenous (IV) infusion (give directly into a vein). In addition, half of the participants will also receive Sigvotatug Vedotin once every 2 weeks as an IV infusion in addition to receiving pembrolizumab.

Participants may receive pembrolizumab for up to about two years. Those participants taking Sigvotatug Vedotin can continue until their NSCLC is no longer responding. The study team will monitorsee how each participant is doing with the study treatment during regular visits at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must meet the following criteria:

   1. Have pathologically confirmed Stage IIIB or IIIC NSCLC and not be a candidate for surgical resection or definitive chemoradiation, or Stage IV NSCLC per the AJCC Staging Manual (Version 8.0) and the UICC Staging System (Eighth edition).
   2. Participants with non-squamous histology must have documented negative test results for EGFR, ALK, and ROS1 AGAs and no known AGAs in NTRK, BRAF, RET, MET, or other AGAs with approved front-line therapies per local standard of care.
   3. Large cell neuroendocrine carcinoma is excluded.
   4. Candidate for treatment with pembrolizumab monotherapy per local guidelines.
2. Tumor has PD-L1 expression in ≥50% of tumor cells (TPS ≥50%) as determined by local testing
3. Measurable disease based on RECIST v1.1 per investigator.
4. Resolution of acute effects of any prior therapy to either baseline severity or NCI CTCAE Grade 1 or less (except for AEs not constituting a safety risk in the investigator's judgment), unless otherwise excluded.

Exclusion Criteria:

1. Life expectancy of <3 months in the opinion of the investigator.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or make the participant inappropriate for the study.
3. Participants with any history of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
4. Known or suspected hypersensitivity, intolerance, or contraindication to any excipient contained in the drug formulation of sigvotatug vedotin or pembrolizumab.
5. Participants with any of the following respiratory conditions:

   1. Evidence of noninfectious or drug-induced ILD or pneumonitis
   2. Known DLCO (adjusted for hemoglobin) <50% predicted.
   3. Grade ≥3 pulmonary disease unrelated to underlying malignancy
6. Known active CNS lesions are excluded. Participants with definitively treated brain metastases (surgery and/or radiotherapy) may be eligible. Clinically inactive brain metastases of longest diameter <0.5 cm are permitted.
7. Major surgery (defined as a surgery requiring inpatient hospitalization of at least 48 hours) within 21 days or minor surgery within 7 days prior to first dose of study intervention.
8. Receipt of a live vaccine within 30 days prior to first dose of study intervention.
9. Pre-existing peripheral neuropathy Grade ≥2 per NCI CTCAE v5.0.
10. Uncontrolled diabetes mellitus, defined as HbA1c ≥8.0% or HbA1c between 7.0% and 8.0% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
11. Prior immune-related AE that led to anti-PD-(L)1 treatment discontinuation, required a high-dose steroid taper (≥0.5 mg/kg prednisone or equivalent per day) for >2 weeks, or required treatment with systemic immunosuppressive therapy.
12. History of autoimmune disease that has required systemic treatment in the past 2 years
13. Participants with prior solid organ or bone marrow transplantation.
14. Currently receiving a high-dose steroid (>10 mg prednisone or equivalent per day) or other immune suppressant or has a condition requiring a chronic high-dose steroid or immune suppressant.
15. Prior and concomitant therapy:

    1. Any prior treatment with MMAE-derived drugs or IB6 targeting agents.
    2. Prior systemic therapy, including anti-PD-(L)1 therapy, for locally advanced, unresectable, or metastatic NSCLC.

       * (Neo)adjuvant anti-PD-(L)1 is allowed if recurrence or progression occurred ≥9 months after the last dose.
       * Other (neo)adjuvant or definitive therapy is allowed if recurrence or progression occurred ≥6 months after the last dose.
    3. Prior radiotherapy to the lung within 6 months of first dose of study intervention, referencing the last date radiotherapy was received.
    4. Chemotherapy, biologics, and/or other antitumor treatment with immunotherapy not specifically prohibited that is completed less than 4 weeks prior to first dose of study intervention, or 2 weeks for palliative radiotherapy.
    5. Any prior therapy with an immune-oncology agent directed to a stimulatory or co-inhibitory T-cell receptor
16. History of or current ongoing infection, including participants positive for active HIV, HBV, or HCV.
17. Severe uncontrolled cardiac or cerebrovascular condition within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2028-09-05 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Baseline to date of death from any cause (Approximately 2 years)
  Overall survival defined as the duration from enrollment to death.
Progression Free Survival (PFS) assessed by blinded independent central review (BICR) | From Baseline to to date of first documentation of progression OR death (Approximately 2 year)
  Progression-free survival is defined as the time interval from the date of randomization to the date of first documented tumor progression determined by blinded independent central review (BICR) assessment as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or death due to any cause, whichever come first.

SECONDARY OUTCOMES:
Progression Free Survival as assessed by Investigator | From Baseline to date of first progression or death (Approximately 4 Years)
  Progression Free Survival (PFS) is defined as the time from the date of first dose of study interventions to the date of first documentation of PD or death due to any cause, whichever occurs first.
Objective Response Rate as assessed by BICR | From Baseline to to the date of progression OR death (approximately to 4 years)
  Objective response rate is defined as the proportion of participants who have a confirmed CR or PR, as best overall response assessed by BICR as per RECIST 1.1, from the date of randomization to the date of disease progression, death due to any cause, whichever occurs first.
Objective Response Rate as assessed by Investigator | From Baseline to to the date of progression OR death (approximately to 4 years)
  defined as the proportion of participants who achieve a best response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Investigator.
Duration of Response as assessed by BICR | From the date of the first objective response to the date of disease progression or death (approximately to 4 years)
  Duration of response is defined as the time from first documented evidence of CR or PR until progressive disease (PD) as determined by BICR assessment as per RECIST 1.1 or death due to any cause, whichever occurs first.
Duration of Response as assessed by Investigator | From the date of the first objective response to the date of disease progression or death (approximately to 4 years)
  defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Number of participants with adverse events (AEs) | From Baseline to end of treatment (up to 4 years)
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Pharmacokinetics (PK) of antibody-conjugated monomethyl auristatin E (ac-MMAE) in plasma: Plasma concentration at end of infusion (CEOI) | Cycle 1 (up to Day 29), Cycle 3 Day 1, Cycle 5 Day 29, Cycle 8 Day 15 and Cycle 11 Day 1
  To characterize the pharmacokinetics (PK) of sigvotatug vedotin when administered in combination with pembrolizumab
PK of ac-MMAE in plasma: Plasma predose concentration (Cpredose) | Cycle 1 (up to Day 29), Cycle 3 Day 1, Cycle 5 Day 29, Cycle 8 Day 15 and Cycle 11 Day 1
  To characterize the pharmacokinetics (PK) of sigvotatug vedotin when administered in combination with pembrolizumab
PK of unconjugated monomethyl auristatin E (MMAE) in plasma: Plasma concentration at end of infusion (CEOI) | Cycle 1 (up to Day 29), Cycle 3 Day 1, Cycle 5 Day 29, Cycle 8 Day 15 and Cycle 11 Day 1
  To characterize the pharmacokinetics (PK) of sigvotatug vedotin when administered in combination with pembrolizumab
PK of MMAE in plasma: Plasma predose concentration (Cpredose) | Cycle 1 (up to Day 29), Cycle 3 Day 1, Cycle 5 Day 29, Cycle 8 Day 15 and Cycle 11 Day 1
  To characterize the pharmacokinetics (PK) of sigvotatug vedotin when administered in combination with pembrolizumab
Number of participants with antidrug antibodies (ADAs) | Cycle 1 (up to Day 29), Cycle 3 Day 1, Cycle 5 Day 29, Cycle 8 Day 15 and Cycle 11 Day 1
  To characterize the immunogenicity of sigvotatug vedotin when administered in combination with pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (240):
- United States (55):
  - Providence St. Jude Medical Center Virginia K. Crosson Cancer Center and Infusion Center, Fullerton, California
  - Providence St. Jude Medical Center, Fullerton, California
  - St. Jude Heritage Medical Group - Fullerton Plaza Multi-Specialty Clinic (Pulmonary Function Test), Fullerton, California
  - Intermountain Health Lutheran Hospital, Golden, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Cancer Centers of Colorado St. Mary's Regional Hospital, Grand Junction, Colorado
  - Intermountain Health St. Mary's Regional Hospital, Grand Junction, Colorado
  - Intermountain Health, Grand Junction, Colorado
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - BRCR Global, Plantation, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Hope and Healing Cancer Services, New Lenox, Illinois
  - Maine Medical Center, Portland, Maine
  - MaineHealth Cancer Care - Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Minnesota Oncology Hematology, PA, Burnsville, Minnesota
  - Minnesota Oncology Hematology PA, Coon Rapids, Minnesota
  - M Health Fairview Cancer Clinic-Edina, Edina, Minnesota
  - Minnesota Oncology Hematology PA, Edina, Minnesota
  - Minnesota Oncology Hematology PA, Fridley, Minnesota
  - Minnesota Oncology Hematology PA, Maple Grove, Minnesota
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology PA, Maplewood, Minnesota
  - Minnesota Oncology Hematology PA, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Health Cancer Center, Robbinsdale, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology, P.A. Cornerstone Medical Specialty Center, Woodbury, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Fremont, Fremont, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Grand Island, Grand Island, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Regional, Grand Island, Nebraska
  - Cancer Partners of Nebraska - April Sampson Cancer Center, Lincoln, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists - Methodist, Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Bergan, Omaha, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Carolina Cancer Research Center, Wilson, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - The University of Texas, MD Anderson Cancer Center - Woodlands, Conroe, Texas
  - Renovatio Clinical - El Paso, El Paso, Texas
  - The University of Texas MD Anderson Cancer Center Diagnostic Imaging, Houston, Texas
  - The University of Texas MD Anderson Cancer Center Investigational Pharmacy Services, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center- Interventional Radiology, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center Clinical Research Imaging, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center - West Houston, Houston, Texas
  - Community Clinical Trials, Kingwood, Texas
  - The University of Texas, MD Anderson Cancer Center - League City, League City, Texas
  - The University of Texas, MD Anderson Cancer Center - Sugar Land, Sugar Land, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Woodlands Radiology, The Woodlands, Texas
  - American Oncology Network Vista Oncology Division-West office, Olympia, Washington
  - American Oncology Network Vista Oncology Division-East office, Olympia, Washington
- Argentina (5):
  - Fundación Respirar, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto Argentino de Diagnóstico y Tratamiento (IADT), Buenos Aires
  - Centro Urológico Profesor Bengió, Córdoba
  - Hospital Privado Universitario de Córdoba, Córdoba
- Australia (5):
  - Campbelltown Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Gympie Hospital, Gympie, Queensland
  - Nambour General Hospital, Nambour, Queensland
- Belgium (5):
  - AZ Sint-Maarten, Mechelen, Antwerpen
  - UZ Brussel, Brussels, Bruxelles-capitale, Région de
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Algemeen Ziekenhuis klina, Brasschaat
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (8):
  - Afecc Associacao Feminina Educacao Combate Cancer, Vitória, Espírito Santo
  - Vencer e Oncoclínica, Teresina, Piauí
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP), Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
- Bulgaria (5):
  - MBAL Uni Hospital, Panagyurishte, Pazardzhik
  - Complex Oncology Center - Burgas, Burgas
  - Medical Center Futuremeds, Plovdiv
  - MHAT for Women's Health Nadezhda, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
- Canada (3):
  - BC Cancer Abbotsford, Abbotsford, British Columbia
  - Centre de Services Ambulatoire de St-Jerome, Saint-Jérôme, Quebec
  - Unité de Recherche Clinique du CISSS des Laurentides, Saint-Jérôme, Quebec
- Chile (7):
  - Clínica Alemana Valdivia, Valdivia, Los Ríos Region
  - Oncocentro Valdivia, Valdivia, Los Ríos Region
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Iceg Clinic, La Florida, Santiago Metropolitan
  - Oncovida, Providencia, Santiago Metropolitan
  - Profar, Providencia, Santiago Metropolitan
  - Clínica Vespucio, Santiago, Santiago Metropolitan
- China (26):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (3):
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice v Motole, Prague, Praha 5
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
- France (15):
  - Centre Antoine-Lacassagne, Nice, Alpes-maritimes
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Centre Hospitalier de Cornouaille Quimper - Concarneau, Quimper, Finistère
  - CHU de Toulouse - Hopital Larrey, Toulouse, Haute-garonne
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-vilaine
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-roussillon
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain, Loire-atlantique
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Val-de-marne
  - Gustave Roussy, Villejuif, Val-de-marne
  - Centre Hospitalier de Cholet, Cholet
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Institut Curie, Paris
- Germany (9):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Klinikum Traunstein, Traunstein, Bavaria
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Klinikum Chemnitz - Flemmingstraße, Chemnitz, Saxony
  - ohO Research GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Labor Berlin, Berlin
  - Vivantes Humboldt Klinikum Apotheke Nord, Berlin
  - Vivantes Hospital Spandau, Berlin
- Greece (8):
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attikí
  - Metropolitan General Hospital, Athens, Attikí
  - Metropolitan Hospital, Athens, Attikí
  - Hygeia Hospital, Marousi, Attikí
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
  - Errikos Dunant Hospital Center, Athens
  - Agios Loukas Clinic, Thessaloniki
- Hungary (2):
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű, Veszprém megye
  - Komárom-Esztergom Vármegyei Szent Borbála Kórház, Tatabánya
- India (4):
  - Spandana Oncology Centre (SOC), Bengaluru, Karnataka
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Venkateshwar Hospital, New Delhi, National Capital Territory of Delhi
- Israel (2):
  - Rabin Medical Center, Petah Tikva, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
- Italy (10):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Istituto Nazionale Tumori Regina Elena, Rome, ROMA
  - Ospedale Isola Tiberina - Gemelli Isola, Rome, ROMA
  - Policlinico "G. Rodolico", Catania, Sicily
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (20):
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Otashi, Gunma
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Mie Chuo Medical Center, Tsu, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - NHO Kinki Chuo Chest Medical Center, Sakai, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka International Cancer Institute, Osaka
- Netherlands (2):
  - Ziekenhuis St. Jansdal, Harderwijk, Gelderland
  - St. Antonius Ziekenhuis, locatie Utrecht, Utrecht
- Poland (6):
  - Med-Polonia Sp. z o. o., Poznan, Greater Poland Voivodeship
  - Instytut Genetyki i Immunologii GENIM, Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandow, Poznan
  - Instytut MSF Sp zoo, Lodz, Łódź Voivodeship
- S C Oncocenter Oncologie Clinica S R L, Timișoara, Timiș County, Romania
- Slovakia (4):
  - Nemocnica AGEL Komarno, Komárno, Nitra Region
  - Fakultna nemocnica Trnava, Trnava, Trnava Region
  - Vychodoslovensky Onkologicky ustav a.s., Košice
  - POKO Poprad s.r.o., Poprad
- South Korea (9):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeonranamdo
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Pusan-kwangyǒkshi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Boramae Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-kwangyǒkshi
- Spain (14):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Dexeus, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Son Llàtzer, Palma, Illes Balears [islas Baleares]
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Quirón Málaga, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
- Inselspital Bern, Bern, Canton of Bern, Switzerland
- Taiwan (8):
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - National Taiwan University Cancer Center (NTUCC), Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Royal Cornwall Hospital, Truro, Cornwall
  - St Bartholomew's Hospital, London, London, CITY of
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Reck M, Lu S, O'Byrne KJ, Barrios C, Pavlov D, Tay F, Negrao MV. Frontline sigvotatug vedotin plus pembrolizumab vs pembrolizumab for non-small cell lung cancer with PD-L1 tumor proportion score >/=50%: phase III study design. Future Oncol. 2025 Dec;21(30):3891-3901. doi: 10.1080/14796694.2025.2596228. Epub 2025 Dec 13. PMID 41388832
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5751003